CLINICAL TRIAL: NCT07100912
Title: A Modified Draize Repeat Insult Patch Test in a Shared Panel of 100 Healthy Volunteers to Investigate the Irritation and Sensitization Potential of 6 Test Articles Following Repeated Cutaneous Patch Applications
Brief Title: Human Skin Safety Testing of 6 Mitopure Topical Products Using a Human Repeat Insult Patch Test (HRIPT) in Healthy Volunteers
Acronym: GLOW-Safety-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Princeton Consumer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ASARIP3M
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Irritation/Irritant; Sensitisation
Keywords: HRIPT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitopure Topical Formula (Experimental)
  Interventions: Other: Mitopure Topical Formula 5; Other: Mitopure Topical Formula 6; Other: Mitopure Topical Formula 7; Other: Mitopure Topical Formula 8; Other: Mitopure Topical Formula 9; Other: Mitopure Topical Formula 10

INTERVENTIONS:
Other: Mitopure Topical Formula 5 — Topical skin cream containing Mitopure
Other: Mitopure Topical Formula 6 — Topical skin cream containing Mitopure
Other: Mitopure Topical Formula 7 — Topical skin cream containing Mitopure
Other: Mitopure Topical Formula 8 — Topical skin serum containing Mitopure
Other: Mitopure Topical Formula 9 — Topical skin exfoliator containing Mitopure
Other: Mitopure Topical Formula 10 — Topical skin cleanser containing Mitopure

SUMMARY:
The objective of this study is to investigate the irritation and sensitization potential of 6 different topically applied test articles containing Mitopure in a shared panel of healthy volunteers by means of repeated cutaneous patch applications under occlusion based on the modified Draize method

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females,18 years of age or older (50% with sensitive skin).
* Completed written informed consent.
* Female subject agrees to use an acceptable method of birth control (e.g. abstinence, condoms, hormonal birth control, IUD, tubal ligation, hysterectomy, bilateral oophorectomy, hysterectomy, post-menopausal for at least one year or male partner vasectomy).

Exclusion Criteria:

* Pregnancy or lactation.
* Participation in a repeat insult patch test (RIPT) or follow-up work within the last month.
* Current treatment by a physician for allergy unless physician consulted by Investigator and participation approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Skin safety as assessed by the number of adverse events of skin irritation and sensitization during human repeat insult patch testing (HRIPT) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- PCR Corp, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No